CLINICAL TRIAL: NCT00305617
Title: Evaluation of CSF Levels of Tarceva (OSI-774) in Patients With Stage III Non-Small Cell Lung Cancer and No CNS Involvement Undergoing Treatment With Tarceva
Brief Title: Cerebrospinal Fluid Levels of Erlotinib in Patients Receiving Erlotinib For Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Diagnostic
Other Study IDs: CASE-CCF-6503; P30CA043703 (NIH); CASE-CCF-6503; CASE-CCF-0967
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2009-07

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Drug Screening Assays, Antitumor

INTERVENTIONS:
Other: antitumor drug screening assay

SUMMARY:
RATIONALE: Determining whether erlotinib passes into the cerebrospinal fluid may help in planning treatment for some types of cancer.

PURPOSE: This clinical trial is studying how well erlotinib is able to pass into the cerebrospinal fluid of patients receiving erlotinib for stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the cerebrospinal fluid penetration of erlotinib in a subset of patients who are undergoing treatment with erlotinib for stage III non-small cell lung cancer and have no CNS metastatic disease.

OUTLINE: This is a pilot, nonrandomized study.

Patients will undergo single lumbar puncture (LP) to remove cerebrospinal fluid for analysis.

After completion of study, patients will be monitored for 1 month after LP to assess for any LP-related complications.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients must be enrolled in the trial: "A Phase I/II Trial of Neoadjuvant Paclitaxel, Carboplatin and OSI-774 (Tarceva) with Concurrent Accelerated Hyperfractionation Radiation Followed by Maintenance Therapy with OSI-774 for Stage III Non-Small Cell Lung Cancer," Principal Investigator: T. Mekhail, M.D.

  * Patient must be in maintenance therapy phase of the study and have received erlotinib for ≥ 1 week
* No known CNS primary or metastatic cancer at any time prior to time of enrollment
* No MRI evidence of pathological enhancement at the time of study entry

PATIENT CHARACTERISTICS:

* Patients must use adequate birth control measures while in the study
* No significant side effects to erlotinib that require dose reduction or interruption
* None of the following medical issues which could make a lumbar puncture unsafe:

  * Platelets < 100,000/mm³
  * INR > 1.1
  * Known bleeding dyscrasia
  * Absolute neutrophil count < 1,500/mm³
  * Ongoing systemic bacterial infection

PRIOR CONCURRENT THERAPY:

* Patients on modest or anti-epileptic therapy must be on nonenzyme-inducing drug only, including any of the following:

  * Neurontin
  * Lamictal
  * Depakote, Depakene
  * Felbatol
  * Keppra
  * Gabitril
  * Topimax
  * Zonegran
* No concurrent enzyme-inducing anti-epileptic drugs such as phenytoin, carbamazepine, or phenobarbital
* No concurrent other drug known to affect the metabolism of erlotinib
* No concurrent anticoagulant therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
CSF penetration as measured by CSF fluid via lumbar puncture on day 7 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Vogelbaum, MD, PhD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States